CLINICAL TRIAL: NCT00352131
Title: A Phase I Study to Assess the Safety and Pharmacokinetics of huC242-DM4 Administered as a Single Intravenous Infusion Once Every Three Weeks to Subjects With Solid Tumors
Brief Title: Maytansinoid DM4-Conjugated Humanized Monoclonal Antibody huC242 in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Clinical Operations, ImmunoGen, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000491224; IMMUNO-101; IMMUNO-045-5011-228; UTHSC-IDD-0504; NCT00625716 (obsolete NCT alias)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Non-colorectal Cancer; Pancreatic Cancer
Keywords: unspecified adult solid tumor, protocol specific; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

INTERVENTIONS:
Drug: HuC242-DM4 — Dose escalation study to define maximum tolerated dose. Doses will vary per cohort. Patients will receive an IV infusion once every three weeks.
  Other Names: IMGN242

SUMMARY:
RATIONALE: Monoclonal antibodies, such as maytansinoid DM4-conjugated humanized monoclonal antibody huC242, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase I trial is studying the side effects and best dose of maytansinoid DM4-conjugated humanized monoclonal antibody huC242 in treating patients with solid tumors that cannot be removed by surgery or have spread to other parts of the body.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and maximum tolerated dose of maytansinoid DM4-conjugated humanized monoclonal antibody huC242 in patients with inoperable or metastatic colorectal cancer, pancreatic cancer, or other solid tumors.

Secondary

* Determine the qualitative and quantitative toxicities of this drug in these patients.
* Characterize the pharmacokinetics of this drug in these patients.
* Describe any antitumor activity of this drug in these patients.

OUTLINE: This is an open-label, nonrandomized, dose-escalation study.

Patients receive maytansinoid DM4-conjugated humanized monoclonal antibody huC242 IV over 4-5 hours on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of maytansinoid DM4-conjugated humanized monoclonal antibody huC242 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Up to 15 patients are treated at the MTD.

Patients undergo blood collection at baseline and periodically during study for pharmacokinetic studies.

After completion of study treatment, patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Inoperable or metastatic disease
* Failed standard therapy
* Confirmed cancer antigen (CanAg) expression

  * Patients must have non-colorectal cancer or pancreatic cancer
  * Tumor must have a homogeneous pattern (i.e., staining present in > 75% of tumor cells for CanAg) and are 2+ or 3+ intensity by immunohistochemistry * No known leptomeningeal disease or progressive brain disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin ≥ 9 g/dL (transfusion allowed)
* Platelet count ≥ 100,000/mm³
* aPTT and INR ≤ 1.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 60 mL/min
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT < 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment
* No hypersensitivity to agents of the same class as the study drug, humanized or nonhumanized antibodies, or immunoconjugates
* No active, uncontrolled infection
* No hepatitis B surface antigen or hepatitis C antibody positivity
* No history of alcoholic liver disease
* No serious medical or psychiatric disorder that would preclude compliance with study requirements
* No peripheral neuropathy > grade 1
* No other malignancy within the past 2 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage A low-grade prostate cancer
* No severe concurrent disease or condition that, in the opinion of the investigator, would preclude study participation

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin C)
* At least 4 weeks since prior radiotherapy, immunotherapy, or hormone therapy for cancer
* At least 4 weeks since prior major surgery
* No concurrent chemotherapy, other immunotherapy, radiotherapy, or other investigational therapy

  * Palliative radiotherapy for related bone metastases allowed
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | for the duration of the trial
Maximum tolerated dose | for the duration of the trial

SECONDARY OUTCOMES:
Toxicity | for the duration of the trial
Pharmacokinetics | for the duration of the trial
Antitumor activity | for the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Alain Mita, MD, Study Chair — Institute for Drug Development
Locations (2):
- United States (2):
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - UT Health Science Center, San Antonio, Texas

REFERENCES:
- [Result] Sankhala KK, Mita AC, Ricart AD, et al.: A phase I and pharmacokinetic study of a CanAg-targeted immunoconjugate, HuC242-DM4, in patients with CanAg-expressing solid tumors. [Abstract] American Association for Cancer Research: Molecular Targets and Cancer Therapeutics, October 22-26, 2007, San Francisco, CA A-B70, 2007.